Study: IMMA-006-14F NCT02530996

4/19/2016

Systemic Sclerosis (SSc) Vasculopathy: Improved Clinical Monitoring and Treatment Statistical analysis

Power calculations were performed using G\*Power computer software version 3. The α-level used for power analysis was set at 0.05. Sample-size calculations were based on the number of patients needed to detect significant differences in FMD between placebo and BH4 (20, 21). With 12 patients/group we had >95% power to detect differences in FMD between placebo and BH4. Statistics were performed using SPSS software (IBM, Chicago, IL). Paired t-tests were used to identify significant changes in measured variables between placebo and BH4. To determine if an effect of visit order was present, the difference in BH4 vs. placebo was calculated and patients were separated into groups based on order of conditions. Unpaired t-tests were used to identify significant changes in measured variables between ordered groups. Statistical significance was set at P<0.05 for all analyses. Data are presented as mean±SEM.